CLINICAL TRIAL: NCT04255277
Title: A Single-center, Double-blind for Cenerimod, Open-label for Moxifloxacin, Placebo-controlled, Parallel-group, Randomized Study in Healthy Male and Female Subjects to Investigate I: the Effect of Cenerimod on the QTc Interval II: the Effect of Cenerimod on the Pharmacokinetics of Combined Oral Contraceptives III: the Effect of Charcoal on the Pharmacokinetics of Cenerimod.
Brief Title: To Study the Effect of Cenerimod on the Electrical Activity of the Heart, in Men and Women. To Study the Effect of Cenerimod on the Use of Oral Contraceptives in Women. To Study the Effect That Charcoal Has on the Elimination of Cenerimod From the Body, in Women and Men.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-064-105; 2019-003156-36 (EudraCT Number)
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Contraceptives, Oral, Combined; Levonorgestrel; Ethinyl Estradiol; Moxifloxacin; cenerimod; Charcoal

STUDY DESIGN:
Intervention Model Description: Period 1: Pharmacokinetic study, Period 2: Thorough-QT and Drug-drug-interaction study. Period 3: Accelerated elimination study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Thorough QT/QTc prolongation (TQT) study is a double-blind parallel study. The accelerated elimination and the combined oral contraceptive pharmacokinetic drug-drug-interaction are open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Period 1: First administration of combined oral contraceptives (Other): Participants randomized to placebo or cenerimod will receive a single oral dose of levonorgestrel (100 μg) and ethinylestradiol (20 μg) in the morning on Day 1.
  Interventions: Drug: Combined oral contraceptives (COC)
- Period 2: Second administration of Combined Oral Contraceptive (Other): Participants randomized to placebo or cenerimod will receive a single oral dose of levonorgestrel (100 μg) and ethinylestradiol (20 μg) in the morning on Day 42.
  Interventions: Drug: Combined oral contraceptives (COC); Drug: Cenerimod 0.5 mg; Drug: Cenerimod 4 mg
- Period 2: Cenerimod 0.5 mg (Experimental): Participants randomized to cenerimod 0.5 mg will receive a single oral dose in the morning from Day 7 to Day 56.
  Interventions: Drug: Combined oral contraceptives (COC)
- Period 2: Cenerimod 4 mg (Experimental): Participants randomized to cenerimod 4 mg will receive a single oral dose in the morning from Day 7 to Day 56.
  Interventions: Drug: Combined oral contraceptives (COC)
- Period 2: Moxifloxacin (Other): Participants randomized to moxifloxacin will receive a single oral 400 mg dose in the morning of Day 42.
  Interventions: Drug: Moxifloxacin 400mg
- Period 2: Placebo (Placebo Comparator): Participants randomized to placebo will receive a single oral dose of placebo in the morning from Day 7 to Day 56.
  Interventions: Drug: Matching Placebo
- Period 3: Cenerimod 0.5 mg and charcoal (Experimental): Participants randomized to cenerimod 0.5 mg in Period 2 will receive 50 g of activated charcoal every 12 hours from Day 57 to Day 67.
  Interventions: Drug: Cenerimod 0.5 mg; Other: Charcoal, activated
- Period 3: Cenerimod 4 mg and charcoal (Experimental): Participants randomized to cenerimod 4 mg in Period 2 will receive 50 g of activated charcoal every 12 hours from Day 57 to Day 67.
  Interventions: Drug: Cenerimod 4 mg; Other: Charcoal, activated
- Period 3: Cenerimod elimination period (No Intervention): Participants randomized to cenerimod 0.5 mg or 4 mg in Period 2 will receive no treatment (i.e., activated charcoal from Day 57 to Day 67) but will have blood samples taken.

INTERVENTIONS:
Drug: Combined oral contraceptives (COC) — A commercially available COC consisting of 0.1mg levonorgestrel and 0.02 mg ethinylestradiol will be used and administered open-label.
  Other Names: Levonorgestrel/Ethinylestradiol
  Arms: Period 1: First administration of combined oral contraceptives; Period 2: Cenerimod 0.5 mg; Period 2: Cenerimod 4 mg; Period 2: Second administration of Combined Oral Contraceptive
Drug: Moxifloxacin 400mg — A commercially available formulation of moxifloxacin 400 mg will be used and administered open-label. All tablets will be from the same batch.
  Arms: Period 2: Moxifloxacin
Drug: Cenerimod 0.5 mg — This will be administered orally as a film-coated tablet in the morning.
  Other Names: ACT-334441
  Arms: Period 2: Second administration of Combined Oral Contraceptive; Period 3: Cenerimod 0.5 mg and charcoal
Drug: Cenerimod 4 mg — This will be administered orally as a film-coated tablet in the morning.
  Other Names: ACT-334441
  Arms: Period 2: Second administration of Combined Oral Contraceptive; Period 3: Cenerimod 4 mg and charcoal
Other: Charcoal, activated — Granules for oral suspension will be used and administered open-label.
  Other Names: Carbomix 50g
  Arms: Period 3: Cenerimod 0.5 mg and charcoal; Period 3: Cenerimod 4 mg and charcoal
Drug: Matching Placebo — Cenerimod matching placebo tablets will be administered once daily orally in the morning.
  Arms: Period 2: Placebo

SUMMARY:
This is a single-center, randomized, double-blind for cenerimod, open-label for moxifloxacin, placebo- and moxifloxacin-controlled, parallel-group study to investigate the effect of cenerimod on the duration of the QT interval in healthy male and female participants.

Participants will be randomly assigned to one of the 4 treatments: placebo, cenerimod 0.5 mg, cenerimod 4 mg or moxifloxacin.

DETAILED DESCRIPTION:
Participants randomized in one of the cenerimod or placebo groups will receive combined oral contraceptives on Day 1 (i.e., prior to cenerimod or placebo administration, Period 1) and on Day 42 (i.e., 36 days after the stat of cenerimod or placebo, Period 2).

Half of the participants randomized in one of the cenerimod or placebo groups will be enrolled in an accelerated elimination procedure part (Period 3).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Body mass index of 18.0 to 29.9 kg/m^2 (inclusive) at the screening.
* No clinically relevant findings on the physical examination at screening.
* Systolic blood pressure 90 to 145 mmHg, diastolic blood pressure 45 to 90 mmHg, and pulse rate 50 to 100 bpm (inclusive), measured on the same arm, after 5 min in the supine position at screening and on Day -1.
* 12-lead ECG without clinically relevant abnormalities, measured after 5 min in the supine position at screening and on admission.
* No clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis) at screening and on admission.
* Negative results from urine drug screen and breath alcohol tests at screening and on admission.
* Women of non-childbearing potential (i.e., postmenopausal [defined as 12 consecutive months with no menses without an alternative medical cause, confirmed by a follicle-stimulating hormone test], with previous bilateral salpingectomy, bilateral salpingo-oophorectomy or hysterectomy, or with premature ovarian failure [confirmed by a specialist]).
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. They must consistently and correctly use (from screening, during the entire study, and up to end-of-study) a highly effective method of contraception with a failure rate of less than 1% per year (i.e., intrauterine device, bilateral tubal occlusion) or be sexually inactive, or have a vasectomized partner. Hormonal contraceptive must not be used within 3 months prior to screening until end of study visit.

Exclusion Criteria:

* Previous exposure to cenerimod.
* Previous exposure to combined oral contraceptive(s), moxifloxacin, or charcoal within 3 months prior to screening.
* Known hypersensitivity to treatments of the same class as cenerimod, or any of the excipients.
* Known hypersensitivity to combined oral contraceptive(s), moxifloxacin, or charcoal or treatments of the same class, or any of their excipients.
* Any contraindication to combined oral contraceptive(s) or moxifloxacin treatment.
* Known hypersensitivity or allergy to natural rubber latex.
* Lymphopenia (< 1000 cells/μL) at Screening and on Day -1.
* Familial history of sick-sinus syndrome.
* Any cardiac condition or illness (including ECG abnormalities) with a potential to increase the cardiac risk of the subject based on the standard 12-lead ECG at screening.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation.
* Clinically relevant history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Any immunosuppressive treatment within 6 weeks or 5 terminal half-lives (t½), whichever is longer, before first study drug administration.
* History or clinical evidence of alcoholism or drug abuse.
* Excessive caffeine consumption, defined as 800 mg or more per day at screening.
* Nicotine consumption within 3 months prior to screening and inability to refrain from nicotine consumption.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals).
* Viral, fungal, bacterial or protozoal infection and / or serology.
* History of deep vein thrombophlebitis or thromboembolic disorders.
* Legal incapacity or limited legal capacity at screening.
* Pregnant or lactating women.
* History or presence of rhythm disorders (e.g., sinoatrial heart block, sick-sinus syndrome, second- or third-degree atrioventricular block, long QT syndrome, symptomatic bradycardia, atrial flutter, or atrial fibrillation) .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected, change-from-baseline QTcF (ΔΔQTcF) | Day 6, 7, 14, 21, 35, and 56.
  ECG variables will be assessed from ECGs extracted in replicates at predefined time points from continuous 24 hour Holter ECG recordings.
Maximum plasma concentration (Cmax): levonorgestrel | Day 1 to Day 3; Day 42 to Day 44
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
Maximum plasma concentration (Cmax): ethinylestradiol | Day 1 to Day 3; Day 42 to Day 44
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
Time to reach Cmax (tmax): levonorgestrel | Day 1 to Day 3; Day 42 to Day 44
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
Time to reach Cmax (tmax): ethinylestradiol | Day 1 to Day 3; Day 42 to Day 44
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
The area under the plasma concentration-time curve (AUC) from zero to infinity (AUC0-inf): levonorgestrel | Day 1 to Day 3; Day 42 to Day 44
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
The area under the plasma concentration-time curve (AUC) from zero to t (AUC0-t): levonorgestrel | Day 1 to Day 3; Day 42 to Day 44
  Blood samples for determination of PK parameters will be collected at predefined
The area under the plasma concentration-time curve (AUC) from zero to infinity (AUC0-inf): ethinylestradiol | Day 1 to Day 3; Day 42 to Day 44
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
The area under the plasma concentration-time curve (AUC) from zero to t (AUC0-t): ethinylestradiol | Day 1 to Day 3; Day 42 to Day 44
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
Terminal elimination half-life (t1/2): levonorgestrel | Day 56 to Day 68
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
Terminal elimination half-life (t1/2): ethinylestradiol | Day 56 to Day 68
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
Terminal elimination half-life (t1/2): cenerimod | Day 56 to Day 68
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
Area under the plasma concentration-time curve (AUC) from Day 56 to infinity (AUC56-inf) for cenerimod | Day 56 to Day 68
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.

SECONDARY OUTCOMES:
Change from baseline in total lymphocyte count to each time point | Day 5, Day 7, Day 14, Day 21, Day 35, Day 56, Day 57, Day 58, Day 1, Day 64, and Day 67
  Blood samples (fasting) collected at predefined time points as part of the normal hematology analysis.
Maximum plasma concentration (Cmax): cenerimod | Day 7, Day 14, Day 21, Day 35, and Day 56
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.
Time to reach Cmax (tmax): cenerimod | Day 7, Day 14, Day 21, Day 35, and Day 56
  Blood samples for determination of pharmacokinetic parameters will be collected at multiple predefined time points.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- Site 1, Rennes, France

IPD SHARING:
Plan to Share IPD: No